CLINICAL TRIAL: NCT06263517
Title: Adaptative, Multicenter, Randomized, Double-blind, Parallel-group, Placebo Controlled, Clinical Trial, on the Efficacy and Tolerability of Different Escalating Doses of Intra-articular Clodronate in Patients With Painful Knee Osteoarthritis
Brief Title: Clinical Trial to Assess Efficacy, Tolerability of Rising Doses of Clodronate in Painful Knee Osteoarthritis Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SPA Società Prodotti Antibiotici S.p.A. (Industry)
Collaborators: Pharmaceutical Development and Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPA-S-899-01-21; 2021-003124-33 (EudraCT Number)
Record Dates: First submitted 2024-01-30; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of Knee
Keywords: Osteoarthritis; Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Clodronic Acid

STUDY DESIGN:
Intervention Model Description: Adaptative, multicenter, randomized, double-blind, parallel-group, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization list will be performed with Proc Plan procedure by SAS ® Software (release 9.4 or later) software using the block randomization method with block size of 4.
  Subjects eligible at Baseline will be randomly allocated to receive 2, 5, 10 /2ml or placebo according to the balanced randomization list.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Intra articular clodronate 2 mg/2 ml once a week for 4 weeks (total clodronate dose = 8 mg)
  Interventions: Drug: Clodronate
- Arm 2 (Experimental): Intra articular clodronate 5 mg/2 ml once a week for 4 weeks (total clodronate dose = 20 mg).
  Interventions: Drug: Clodronate
- Arm 3 (Experimental): Intra articular clodronate 10 mg/2 ml once a week for 4 weeks (total clodronate dose = 40 mg)
  Interventions: Drug: Clodronate
- Arm 4 (Placebo Comparator): Placebo 2 ml once a week for 4 weeks (total clodronate dose = 0 mg).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clodronate — For Arm 1, patients will be treated with intra articular clodronate 2 mg/2 ml from Baseline to Week 3
  Arms: Arm 1
Drug: Clodronate — For Arm 2, patients will be treated with intra articular clodronate 5 mg/2 ml from Baseline to Week 3
  Arms: Arm 2
Drug: Clodronate — For Arm 3, patients will be treated with intra articular clodronate 10 mg/2 ml from Baseline to Week 3
  Arms: Arm 3
Drug: Placebo — For Arm 4, patients will be treated with Placebo 2 ml from Baseline to Week 3
  Arms: Arm 4

SUMMARY:
The goal of this clinical trial is to to clarify which is the best dose of administration, to select a dose and to confirm the therapeutic efficacy of clodronate in patients with painful knee osteoarthritis (OA). The clinical trial will be divided in two parts.

The main questions it aims to answer are:

* in Phase II, to assess the safety and tolerability of different escalating doses of intra articular (IA) clodronate
* in Phase II, to set a defined therapeutic dose (DTD) to be used in Phase III
* in Phase III, to assess the safety and tolerability of different escalating doses of IA clodronate to confirm and extensively evaluate the therapeutic efficacy and safety of the clodronate DTD in patients with knee OA

DETAILED DESCRIPTION:
The phase II will be a multicenter, double-blind, randomized, placebo-controlled, parallel group four-arm study, according to the treatment dose (dose finding).

Briefly, 4 groups of 74 patients (in order to have 64 fully evaluated patients taking into consideration 10 patients dropped out), i.e. a total of 296 patients, with knee OA each will be randomly allocated to the following treatments:

1. IA clodronate 2 mg/2 ml once a week for 4 weeks (total clodronate dose = 8 mg).
2. IA clodronate 5 mg/2 ml once a week for 4 weeks (total clodronate dose = 20 mg).
3. IA clodronate 10 mg/2 ml once a week for 4 weeks (total clodronate dose = 40 mg).
4. Placebo 2 ml once a week for 4 weeks (total clodronate dose = 0 mg).

At the end of phase II, the minimum effective clodronate dose will be selected as DTD for the Phase III.

The phase III will be a multicenter, double-blind, randomized, placebo-controlled, two parallel groups (DTD vs. placebo) study.

Briefly, patients with knee OA will be randomly assigned to two experimental groups:

1. the DTD defined during the Phase II.
2. Matching placebo. The sample size of Phase III will be definitively calculated according to the extent of pain Visual Analogue Scale (VAS) reduction observed in the Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged 50 up to 75 years at ICF signature.
* Diagnosis of knee OA according to the American College of Rheumatology, confirmed by Rx during the screening (a Rx performed in the last 3 months before Baseline is accepted).
* Kellgren-Lawrence radiographic score between 2 and 3 degrees in the tibiofemoral joint.
* Symptomatic knee OA (pain) since at least 6 months with a knee pain (VAS) ranging between 40 and 80 mm at Screening visit (the figure should be confirmed at Baseline).
* Female patients of childbearing potential must have a negative pregnancy test before each treat-ment and during the Visit 5 - Week 4 and they must use adequate methods of contraception throughout the course of the study.
* A signed ICF by the patient after exhaustive study discussion with the investigators.

Exclusion Criteria:

* BMI > 35 kg/m² (Class II obesity).
* Joint instability due to other reasons than knee OA, such as f.i. algo dystrophic syndrome, either partial or complete rupture of internal / externals ligaments, kneecap instability, etc.
* Otherwise located lower limb pain, such as hip pain.
* Other musculoskeletal disorders related to the target knee.
* Any treatment with IA drugs in the last 3 months before Day 0 - Baseline (including any formulation of corticosteroids or hyaluronic acid injections).
* Corticosteroid use by any systemic route, and hyaluronic acid injection or intraarticular corticosteroids for any other joint in the previous month will not be permitted.
* Any treatment with systemic non-steroidal anti-inflammatory drugs (NSAIDs) in the week before enrolment, or any steroid anti-inflammatory drugs and chondroprotective drugs in the thirty (30) days before month before Baseline.
* Any treatment with systemic bisphosphonates in the last twelve (12) months before Baseline.
* Any treatment with Glucosamine or Chondroitin sulfate, Diacerein and Matrix metalloproteinase (MMP) inhibitors in the 4 weeks before Baseline.
* Any treatment with Denosumab in the twelve (12) months before Baseline.
* Any treatment with Paracetamol in the twelve (12) hours before Baseline.
* Any knee surgery in the past or knee arthroplasty.
* Any diagnostic or surgical arthroscopy of the knee in the six (6) months before Baseline.
* Any jaw osteonecrosis in the last twenty-four (24) months before Baseline or at a risk of jaw osteonecrosis.
* Any known hypersensitivity to the drug in the study to its excipients or other bisphosphonates, and any hypersensitivity to Paracetamol (rescue drug).
* Any participation in a clinical study in which the last administration of the investigational medicinal product was within two (2) weeks before consenting to study participation (i.e.signing ICF).
* Inadequate organ function defined by the following laboratory parameters:

  1. Absolute Neutrophil Count (ANC) < 1500/μl.
  2. Hemoglobin (Hb) < 9 g/dl (< Hb 5.6 mmol/L)
  3. Platelet Count < 100.000/μl
  4. Serum Creatinine > 1.5 x Upper limit normal (ULN) or estimated Glomerular Filtration Rate (eGFR) < 60 mL/min (as per Cockroft-Gault formula).
  5. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST)> 1.5 x Upper limit normal(ULN).
  6. Serum Total Bilirubin > 1.5 x Upper limit normal (ULN).
* Pregnant or breastfeeding women, or women planning to become pregnant during the study.
* Any positive or suspected history of alcoholism or drug use.
* Clinically significant (i.e.) gastrointestinal, renal, hepatic, pulmonary, cardiovascular or neurological disease that could interfere with the outcome of the study or the patient's ability to comply with study requirements.
* Patients unwilling or unable to comply with the protocol.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy: VAS Reduction | Week 7
  A clodronate dose will be considered as effective when a ≥ 10 mm reduction in the Visual Analogue Scale (VAS) of knee pain will be observed at Week 7 vs. Placebo

SECONDARY OUTCOMES:
VAS mean changes | At Screening, at Baseline, at Weeks 1, 2, 3, 4, 5, 11, 15
  Mean changes in the Visual Analogue Scale (VAS) of knee pain observed at each other visit than Week 7 vs. Placebo and vs Baseline.
VAS mean changes observed 120 minutes after IA | At Baseline and at Weeks 1, 2 and 3
  Mean changes in the Visual Analogue Scale (VAS) of knee pain observed 120 minutes after IA injection at Baseline, Weeks 1, 2 and 3 vs predose assessment
Lequesne Algofunctional Index mean changes | At Screening, at Baseline, at Weeks 1, 2, 3, 4, 5, 7, 11, 15
  Mean changes in the Lequesne Algofunctional Index at each visit vs Placebo and vs Baseline.
WOMAC mean changes | At Screening, at Baseline, at Weeks 1, 2, 3, 4, 5, 7, 11, 15
  Mean changes in the (WOMAC) Western Scale Ontario MacMaster Index at each visit vs Placebo and vs Baseline.
Range of motion mean changes | At Screening, at Baseline, at Weeks 1, 2, 3, 4, 5, 7, 11, 15
  Mean changes in the Range of Motion at each visit vs Placebo and vs Baseline.
Paracetamol consumption | At Baseline, at Weeks 1, 2, 3, 4, 5, 7, 11, 15
  Use of rescue drug consumption (paracetamol) across the patients visits

OTHER OUTCOMES:
SAE Reporting | At Screening, at Baseline, at Weeks 1, 2, 3, 4, 5, 7, 11, 15
  Recording of Serious adverse event (SAE) and abnormal laboratory or any clinical signs of intolerance across the patients' visits.
AE Reporting | At Screening, at Baseline, at Weeks 1, 2, 3, 4, 5, 7, 11, 15
  Recording of adverse event (AE)
Clinical signs of intolerance Recording | At Baseline, at Weeks 1, 2, 3, 4, 5, 7, 11, 15
  Recording of any clinical signs of intolerance across the patients' visits

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - IRCCS Istituti Clinici Maugeri, Castel Goffredo, Mantova
  - Ospedale San Pellegrino, Castiglione delle Stiviere, Mantova
  - Ospedale Civile Servizio di Riabilitazione Funzionale, Volta Mantovana, Mantova
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Centro Riabilitativo Polifunzionale Teresio Borsalino, Alessandria
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Israelitico, Roma
  - Ospedale San Pietro, Rome
  - Ospedale San Paolo, Savona
  - Azienda Ospedaliero Universitaria Senese, Siena
  - Ospedale Policlinico "G.B. Rossi" Borgo Roma, Verona